CLINICAL TRIAL: NCT04501861
Title: Hemodynamic Effect of Norepinephrine Versus Vasopressin on the Pulmonary Circulation in Cardiac Surgery Patients: a Comparative-effectiveness Quality Project
Brief Title: Hemodynamic Effect of Norepinephrine Versus Vasopressin on the Pulmonary Circulation in Cardiac Surgery Patients:
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-301
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases | interventions — Vasopressins; Norepinephrine

STUDY DESIGN:
Intervention Model Description: Randomized cluster crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- use of vasopressin (Active Comparator): Hemodynamic effect of vasopressin on the pulmonary circulation in cardiac surgery patients
  Interventions: Drug: Norepinephrine
- use of norepinephrine (Active Comparator): Hemodynamic effect of norepinephrine on the pulmonary circulation in cardiac surgery patients
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — Vasopressin (20 IU/100 ml in 5% dextrose) were stored in pre-mixed bags in the operating room, readily available for continuous infusion administration via pre-programed infusion pumps
  Arms: use of norepinephrine
Drug: Norepinephrine — Norepinephrine (4 mg/250ml in 5% dextrose) were stored in pre-mixed bags in the operating room, readily available for continuous infusion administration via pre-programed infusion pumps
  Arms: use of vasopressin

SUMMARY:
The relative increase in the mPAP with the same unit increase in MAP adjusted for baseline, and RV function assessed by GLS, between VP and NE in patients with normal and increased pulmonary artery pressure, who require vasopressor support during cardiac surgery.

DETAILED DESCRIPTION:
The specific aims of our study are to compare 1) the relative increase in the mPAP with the same unit increase in MAP adjusted for baseline and 2) RV function assessed by GLS, between VP and NE in patients with normal and increased pulmonary artery pressure, who require vasopressor support during cardiac surgery. We hypothesize that the use of vasopressin compared with norepinephrine induces a lower mPAP-to-MAP ratio, in cardiac surgical patients with and without pulmonary hypertension who require intraoperative vasopressor support. Second, we will test the hypothesis that vasopressin is associated with improved right ventricular global longitudinal strain compared to norepinephrine in patients requiring vasopressor support during cardiac surgery.

ELIGIBILITY:
Inclusion criteria:

Adults> 18 years of age

* Elective cardiac surgery with the use of CPB
* Patients with pulmonary artery catheter insertion
* Systemic hypotension (MAP < 70 mmHg) requiring continuous infusion of vasopressor

Exclusion Criteria:

* Transplant surgery
* Ventricular assist device implantation other than intra-aortic balloon counter-pulsation
* Pulmonary endarterectomy
* Thoracoabdominal aneurysm repair
* Inhalational pulmonary vasodilators (e.g. Epoprostenol) administration before insertion of pulmonary artery catheter
* Vasopressin is started as the first choice of pressor per clinical staff discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariya Geube, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a unblinded alternating trial. The treatment will be randomized in one week blocks and not by patient, using the RedCap system. This means that during any week, eligible patients will be exposed to the same vasopressor agent (vasopressin or norepinephrine). And the following week there will be new randomization in place. Allocations will be directly communicated to anesthesia personnel and by signs prominently displayed in anesthesia ready room.
Groups:
- The Use of Vasopressin: This group including patients who received vasopressin on the pulmonary circulation in cardiac surgery.
- The Use of Norepinephrine: This group including patients who received norepinephrine on the pulmonary circulation in cardiac surgery.
Period: Overall Study
Arm/Group | The Use of Vasopressin | The Use of Norepinephrine
Started | 70 | 83
Completed | 0 | 0
Not Completed | 70 | 83

BASELINE CHARACTERISTICS:
Population: In the final study population, 153 patients were included.
Groups:
- Patients Using Intraoperative Vasopressin: Hemodynamic effect of vasopressin on the pulmonary circulation in cardiac surgery patients
- Patients Using Intraoperative Norepinephrine: Hemodynamic effect of Norepinephrine on the pulmonary circulation in cardiac surgery patients
- Total: Total of all reporting groups
Arm/Group | Patients Using Intraoperative Vasopressin | Patients Using Intraoperative Norepinephrine | Total
Number analyzed (Participants) | 70 | 83 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12) | 66 (13) | 66 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 32 | 50
  Male | 52 | 51 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 70 | 83 | 153
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29 (6) | 28.2 (6.5) | 28.5 (6.5)
Comorbid conditions [Count of Participants; unit: Participants]
  Hypertension | 53 | 66 | 119
  Coronary artery disease | 49 | 61 | 110
  Diabetes | 21 | 29 | 50
  Chronic kidney disease | 2 | 7 | 9
  Peripheral artery disease | 9 | 17 | 26
  Cerebral vascular disease | 12 | 24 | 36
  Congestive heart failure | 30 | 39 | 69
  Smoking history | 34 | 43 | 77
  Hyperlipidemia | 42 | 51 | 93
  Pulmonary hypertension | 19 | 21 | 40
Preoperative RV dysfunction [Count of Participants; unit: Participants] — Right Ventricular (RV) Dysfunction refers to the impaired function of the right ventricle of the heart, which is responsible for pumping deoxygenated blood from the body into the lungs for oxygenation. RV dysfunction can lead to inadequate blood flow to the lungs and subsequent systemic complications.
  Participants
    Normal | 50 | 63 | 113
    Mild | 14 | 14 | 28
    Moderate or severe | 6 | 6 | 12
Surgery type [Count of Participants; unit: Participants]
  Aortic valve surgery | 13 | 8 | 21
  Aortic surgery | 7 | 5 | 12
  CABG + aortic valve surgery | 9 | 7 | 16
  CABG + mitral valve surgery | 3 | 4 | 7
  Isolated CABG | 10 | 15 | 25
  Mitral valve surgery | 4 | 8 | 12
  Multi-valve procedures | 18 | 33 | 51
  Other | 6 | 3 | 9
Primary or repeat surgery [Count of Participants; unit: Participants]
  Primary surgery | 38 | 50 | 88
  Reoperative surgery | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: mPAP-to-MAP Ratio
Description: The intraoperative mean pulmonary artery pressure(mPAP) adjusted for systemic mean arterial pressure(MAP), using a time-weighted average mPAP-to-MAP ratio measured during 20 minute period after chest closure
Time Frame: during 20 minute period after chest closure
Population: Not all the patients in the 2 groups with preoperative pulmonary arterial hypertension, we only included the eligible patients.
Measure: Mean (Standard Deviation); unit: ratio of mPAP-to-MAP
Groups:
- The Use of Vasopressin: Vasopressin (20 IU/100 ml in 5% dextrose) was stored in pre-mixed bags in the operating room, readily available for continuous infusion administration via pre-programed infusion pumps
  Hemodynamic effect of vasopressin on the pulmonary circulation in cardiac surgery patients
- The Use of Norepinephrine: Norepinephrine (4 mg/250ml in 5% dextrose) was stored in pre-mixed bags in the operating room, readily available for continuous infusion administration via pre-programed infusion pumps
  Hemodynamic effect of norepinephrine on the pulmonary circulation in cardiac surgery patients
Arm/Group | The Use of Vasopressin | The Use of Norepinephrine
Number analyzed (Participants) | 70 | 83
ratio of mPAP-to-MAP
  mPAP-to-MAP ratio | 0.394 (0.086) | 0.385 (0.094)
  mPAP-to-MAP ratio with preop pulmonary hypertension: number analyzed (Participants) | 40 | 52
  mPAP-to-MAP ratio with preop pulmonary hypertension | 0.42 (0.082) | 0.40 (0.093)
  mPAP-to-MAP ratio without preop pulmonary hypertension: number analyzed (Participants) | 29 | 31
  mPAP-to-MAP ratio without preop pulmonary hypertension | 0.37 (0.084) | 0.36 (0.092)
Statistical Analysis 1: Comparison: The Use of Vasopressin vs The Use of Norepinephrine; Test type: Equivalence — Compare mPAP-to-MAP ratio between patients who received norepinephrine versus vasopressin intraoperatively. Post intervention measurements will be recorded after protamine administration until end of chest closure; p = 0.53, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.043 to 0.022]
Statistical Analysis 2: Comparison: The Use of Vasopressin vs The Use of Norepinephrine; mPAP-to-MAP ratio was compared between patients with pre-existing pulmonary hypertension of use of vasopressin and norepinephrine. Preoperative pulmonary arterial hypertension was defined by using the cut-off value of 25 mmHg for the time-weighted average mPAP, i.e., time weighted average mPAP < 25 mmHg indicated absence of preoperative pulmonary arterial hypertension; otherwise, presence of preoperative pulmonary hypertension; Test type: Equivalence — Compare mPAP-to-MAP ratio between patients who with preop PH received norepinephrine versus vasopressin intraoperatively. Post intervention measurements will be recorded after protamine administration until end of chest closure. The number of patients in norepinephrine group is 52 and in vasopressin group is 40. The significance level was 0.05 for all analyses. All tests were 2-sided. Interactions were considered significant when the interaction P was < 0.10; p = 0.26, Mixed Models Analysis; Mean Difference (Final Values) = -0.022, 95% CI 2-sided [-0.061 to 0.016]
Statistical Analysis 3: Comparison: The Use of Vasopressin vs The Use of Norepinephrine; mPAP-to-MAP ratio was compared between patients without pre-existing pulmonary hypertension of use of vasopressin and norepinephrine. Preoperative pulmonary arterial hypertension was defined by using the cut-off value of 25 mmHg for the time-weighted average mPAP, i.e., time weighted average mPAP < 25 mmHg indicated absence of preoperative pulmonary arterial hypertension; otherwise, presence of preoperative pulmonary hypertension; Test type: Equivalence — Compare mPAP-to-MAP ratio between patients who without preop PH received norepinephrine versus vasopressin intraoperatively. Post intervention measurements will be recorded after protamine administration until end of chest closure. The number of patients in norepinephrine group is 31 and in vasopressin group is 29. The significance level was 0.05 for all analyses. All tests were 2-sided. Interactions were considered significant when the interaction P was < 0.10; p = 0.88, Mixed Models Analysis; Mean Difference (Final Values) = -0.0035, 95% CI 2-sided [-0.05 to 0.043]

2. Secondary Outcome: RV Free Wall Strain
Description: Right Ventricular Free Wall Longitudinal Strain (RV FWLS) is a measure of the deformation (strain) of the right ventricle's free wall (the part not attached to the septum) during contraction. It quantifies how much the myocardium in the free wall of the right ventricle shortens along its longitudinal axis (base to apex) during systole (contraction). It is expressed as a negative percentage (%), where more negative values indicate better contractility (e.g., -20% is better than -10%). In this study, it was measured by transesophageal echocardiography in the 2D mid-esophageal four-chamber view during a steady state period after chest closure
Time Frame: during 20 minutes period after chest closure
Population: Included all patients for RV free wall strain. As not all the patients with/without preoperative pulmonary arterial hypertension, so the study pop in subgroup are different.
Measure: Mean (Standard Deviation); unit: percentage of RV free wall strain
Groups:
- The Use of Vasopressin: Vasopressin (20 IU/100 ml in 5% dextrose) were stored in pre-mixed bags in the operating room, readily available for continuous infusion administration via pre-programed infusion pumps.
  Hemodynamic effect of vasopressin on the pulmonary circulation in cardiac surgery patients
- The Use of Norepinephrine: Norepinephrine (4 mg/250ml in 5% dextrose) was stored in pre-mixed bags in the operating room, readily available for continuous infusion administration via pre-programed infusion pumps.
  Hemodynamic effect of norepinephrine on the pulmonary circulation in cardiac surgery patients
Arm/Group | The Use of Vasopressin | The Use of Norepinephrine
Number analyzed (Participants) | 70 | 83
percentage of RV free wall strain
  RV free wall strain | -18.2 (8.4) | -19.4 (7.2)
  RV free wall strain with preop pulmonary hypertension: number analyzed (Participants) | 28 | 34
  RV free wall strain with preop pulmonary hypertension | -17.5 (8.4) | -18.9 (8.1)
  RV free wall strain without preop pulmonary hypertension: number analyzed (Participants) | 18 | 22
  RV free wall strain without preop pulmonary hypertension | -19.2 (8.4) | -20.0 (5.7)
Statistical Analysis 1: Comparison: The Use of Vasopressin; Test type: Equivalence — Imbalanced confounders such as female, coronary artery disease, preoperative ejection fraction, surgery type, primary or repeat surgery, and bypass time were additionally adjusted. A different inverse probability of treatment weighting was fit for secondary analysis and a linear mixed regression model with random intercept to account for intra-week correlation to estimate the effect of norepinephrine on right ventricular free wall strain using the new obtained stabilized weights; p = 0.37, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-6.0 to 2.3]
Statistical Analysis 2: Comparison: The Use of Vasopressin vs The Use of Norepinephrine; RV free wall strain compare between patients with pre-existing pulmonary hypertension of use of vasopressin and norepinephrine. Preoperative pulmonary arterial hypertension was defined by using the cut-off value of 25 mmHg for the time-weighted average mPAP, i.e., time weighted average mPAP < 25 mmHg indicated absence of preoperative pulmonary arterial hypertension; otherwise, presence of preoperative pulmonary hypertension;; Test type: Equivalence — We examined the effect of norepinephrine versus vasopressin on right ventricular free wall strain by considering patients who have preoperative pulmonary hypertension. The number of patients in norepinephrine group is 34 and in vasopressin group is 28. The significance level was 0.05 for all analyses. All tests were 2-sided. The significance levels of subgroup analyses were not corrected for multiple comparisons. Interactions were considered significant when the interaction P was < 0.10; p = 0.39, Mixed Models Analysis; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-7.1 to 2.8]
Statistical Analysis 3: Comparison: The Use of Vasopressin vs The Use of Norepinephrine; We examined the effect of norepinephrine versus vasopressin on right ventricular free wall strain by separately considering patients who did not have preoperative pulmonary hypertension. Preoperative pulmonary arterial hypertension was defined by using the cut-off value of 25 mmHg for the time-weighted average mPAP, i.e., time weighted average mPAP < 25 mmHg indicated absence of preoperative pulmonary arterial hypertension; otherwise, presence of preoperative pulmonary hypertension; Test type: Equivalence — We're going to explore the interaction between preoperative pulmonary arterial hypertension status and treatment group by equivalence analysis. The number of patients in norepinephrine group is 22 and in vasopressin group is 18.The significance level was 0.05 for all analyses. All tests were 2-sided. The significance levels of subgroup analyses were not corrected for multiple comparisons. Interactions were considered significant when the interaction P was < 0.10; p = 0.63, Mixed Models Analysis; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-7.6 to 4.6]

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- The Use of Vasopressin: Hemodynamic effect of vasopressin on the pulmonary circulation in cardiac surgery patients
- The Use of Norepinephrine: Hemodynamic effect of norepinephrine on the pulmonary circulation in cardiac surgery patients
Arm/Group | The Use of Vasopressin | The Use of Norepinephrine
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Our study protocol excluded patients at particularly high risk for acute right ventricular failure. Thus, our conclusions should not be extrapolated to such vulnerable populations. Our analysis was not adequately powered to evaluate mortality and other major clinical outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT04501861/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT04501861/ICF_001.pdf